CLINICAL TRIAL: NCT05362227
Title: Lower Gastrointestinal Bleeding in the Emergency Department: High-Volume Vs Low-Volume Peg Bowel Preparation for Colonoscopy
Brief Title: High-Volume Vs Low-Volume Preparation in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, OJETTI VERONICA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20192668
Record Dates: First submitted 2022-04-29; First posted 2022-05-05 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: GastroIntestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Volume (Other): Patients in the group were instructed to take 4 L of solution on the day before the colonoscopy
  Interventions: Drug: High volume macrogol
- Low-Volume (Other): Patients in the group were instructed to take 2 L of solution on the day before the colonoscopy
  Interventions: Drug: Low volume macrogol

INTERVENTIONS:
Drug: Low volume macrogol — Clensia 2 lt
  Arms: Low-Volume
Drug: High volume macrogol — Selg 4 lt
  Arms: High-Volume

SUMMARY:
The primary endpoint of this study was to compare the intestinal cleansing of patients with LGIB requiring colonoscopy, prepared with High-Volume or with Low-Volume who have to perform colonoscopy, directly from the ED. The intestinal cleansing was evaluated with the standardized Boston Bowel Preparation Scale (BBPS).

The secondary endpoint was to evaluate the tolerability and compliance of patients prepared with High-Volume in comparison to Low-Volume in the ED.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* > 18 years and <85 years,
* hemodynamically stable,
* able to sign informed consent
* requiring colonoscopy
* anemia (loss of at least 2 g/dl of Hb) with or without active bleeding

Exclusion Criteria:

* suspected or confirmed pregnancy,
* hemodynamically unstable patients,
* patients unable to swallow or with known or suspected gastrointestinal obstruction or perforation,
* toxic megacolon,
* major colonic resection,
* heart failure (Class III or IV NYHA),
* severe liver failure,
* end-stage renal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
intestinal cleansing | during colonscopy procedure
  Using Boston Bowel Preparation Scale score (from 0 to 9, where 9 is worst preparation level)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Ojetti, Prof, Principal Investigator — Fondazione Policlinico universitario a. Gemelli
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saviano A, Petruzziello C, Riccioni ME, Di Pumpo M, Petrucci M, Brigida M, Zanza C, Candelli M, Franceschi F, Ojetti V. Lower Gastrointestinal Bleeding in the Emergency Department: High- Volume vs. Low-Volume Peg Bowel Preparation for Colonoscopy: A Randomized Trial. Rev Recent Clin Trials. 2023;18(1):76-81. doi: 10.2174/1574887117666220908152754. PMID 36089784